CLINICAL TRIAL: NCT05958966
Title: Effects of e-Cigarettes on Perceptions and Behavior - Substudy 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Adam Leventhal, Professor, Department of Preventive Medicine, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: HS-18-00839 Substudy 2
Record Dates: First submitted 2023-07-07; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Electronic Cigarette Use; E-Cig Use; Cigarette Smoking; Cigarette Use, Electronic
MeSH Terms: conditions — Vaping; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- E-cigarette e-liquid 1 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Other: E-cigarette e-liquid self-administration
- E-cigarette e-liquid 2 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Other: E-cigarette e-liquid self-administration
- E-cigarette e-liquid 3 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Other: E-cigarette e-liquid self-administration
- E-cigarette e-liquid 4 (Experimental): Participants will self-administer an e-cigarette e-liquid.
  Interventions: Other: E-cigarette e-liquid self-administration
- No e-liquid (No Intervention): Participants do not receive an e-cigarette e-liquid to self-administer.

INTERVENTIONS:
Other: E-cigarette e-liquid self-administration — Participant will self-administer an experimenter-provided e-cigarette.
  Arms: E-cigarette e-liquid 1; E-cigarette e-liquid 2; E-cigarette e-liquid 3; E-cigarette e-liquid 4

SUMMARY:
This project will assess the ways in which e-cigarette product diversity impacts the user experience to inform potential regulations by identifying product characteristics that may: (1) put young adults at risk for tobacco product use; and (2) facilitate adult smokers switching to e-cigarettes. There are three primary objectives to the study: (1) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect product appeal across young adult e-cigarette users and middle-age/older adult smokers; (2) Determine which dimensions of e-cigarette product diversity differentially affect product appeal in the overall population of tobacco product users as well as affect abuse liability in young adult e-cigarette users and the ability to resist smoking in adult smokers; (3) Determine the affect of product characteristics on e-cigarette nicotine delivery profile. For this substudy, adult smokers (N=200) will attend two laboratory session in which they will self-administer e-cigarette products varied according to within-subject e-cigarette factors (e.g., flavor, nicotine formulation) and smoke their own cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Regular use of cigarettes containing nicotine.

Exclusion Criteria:

* Pregnant or planning to become pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Subjective Appeal Rating Questionnaire | 1 hour
  This self-report measure of product appeal will be completed following e-cigarette self-administration. Scores can range from 0 to 100 for the appeal rating, with lower scores representing lower levels of appeal and higher scores representing higher levels of appeal.
Sensory Attributes Rating Questionnaire | 1 hour
  This self-report measure of product sensory attributes will be completed following e-cigarette self-administration. Scores can range from 0 to 100 for the sensory attribute rating, with lower scores representing lower levels of liking the sensory attribute and higher scores representing greater liking of the sensory attribute.
Smoking Delay Task | 1 hour
  Minutes delayed before purchasing time to smoke own cigarettes. Scores can range from 0mins to 50mins for the smoking delay task, with lower scores representing fewer minutes delayed from smoking and higher scores representing longer minutes delayed from smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No